CLINICAL TRIAL: NCT03350360
Title: Randomized Clinical Trials of Attention Control Training for PTSD Related to Combat or Interpersonal Violence
Brief Title: Attention Control Training for PTSD Related to Combat or Interpersonal Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Amy Badura Brack, Professor of Psychology, Creighton University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1123259
Record Dates: First submitted 2017-11-16; First posted 2017-11-22 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Random assignment and coded entry to a computer website
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention Control Training Clinic (Experimental): Attention Control Training Clinic will consist of:
  * 6 sessions in the clinic lasting approximately 10 minutes each.
  * Each session will consist of 128 presentations of pairs of neutral and threatening stimuli, followed by the presentation of a response cue (right or left arrow to be clicked on a computer keyboard).
  Interventions: Behavioral: Attention Control Training
- Attention Control Training Web-delivery (Experimental): Attention Control Training Web-delivery will consist of:
  * 6 sessions lasting approximately 10 minutes each logged into via the internet from the participants' home.
  * Each session will consist of 128 presentations of pairs of neutral and threatening stimuli, followed by the presentation of a response cue (right or left arrow to be clicked on a computer keyboard).
  * Ideally participants will complete 2 sessions per week, allowing them to complete the trial in less than one month's time
  Interventions: Behavioral: Attention Control Training
- Comparison Task Clinic (Placebo Comparator): * 6 sessions in the clinic of a presumably inactive neutral-neutral stimuli intervention lasting approximately 10 minutes each.
  * Each session will consist of 128 presentations of pairs of faces, followed by the presentation of a response cue (right or left arrow to be clicked on a computer keyboard).
  (Note that those receiving this arm, are invited to repeat the attention control training web-delivery arm at the end of their participation).
  Interventions: Behavioral: Attention Control Training; Behavioral: Comparison Task

INTERVENTIONS:
Behavioral: Attention Control Training — Attention control training teaches participants that the emotional salience of cues (i.e., threatening or neutral) is not related to successful completion of the computerized response task, and thus, teaches participants to ignore irrelevant threat-related contingencies (Badura-Brack et al., 2015).
Behavioral: Comparison Task — Neutral- neutral stimuli prior to response task
  Arms: Comparison Task Clinic

SUMMARY:
Participants will complete a pre and post training psychological assessment. Participants will be assigned to attention control training or the comparison stimuli computer task in a double-blind randomized control trial design. Both computerized dot probe tasks display two stimuli on a computer screen, one above the other, followed by a small right or left arrow appearing in the location vacated by one of the stimuli. Participants are required to respond as quickly as they can by pressing the indicated right or left arrow on their computer keyboard without compromising accuracy. Participants complete 6 training sessions.

ELIGIBILITY:
Inclusion Criteria:

* military veteran or woman exposed to interpersonal violence (e.g. domestic or sexual violence).
* significant symptoms of PTSD

Exclusion Criteria:

* bipolar disorder, schizophrenia, OCD, unable to attend sessions sober.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Change in posttraumatic stress disorder (PTSD) symptoms from pre to post test | 30 minute long administration at both pre and post training to measure change. (repeat assessments are conducted 1 month apart)
  Structured diagnostic interview for PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton University, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badura-Brack AS, Naim R, Ryan TJ, Levy O, Abend R, Khanna MM, McDermott TJ, Pine DS, Bar-Haim Y. Effect of Attention Training on Attention Bias Variability and PTSD Symptoms: Randomized Controlled Trials in Israeli and U.S. Combat Veterans. Am J Psychiatry. 2015 Dec;172(12):1233-41. doi: 10.1176/appi.ajp.2015.14121578. Epub 2015 Jul 24. PMID 26206075

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03350360/Prot_SAP_000.pdf